CLINICAL TRIAL: NCT04807465
Title: How Does Smoking Effect the Clinical Performance of a Universal Adhesive Used With Different Application Modes in Non Carious Cervical Lesions?
Brief Title: Different Modes of Universal Adhesive in Smokers and Non-Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, A Ruya Yazici, professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: interventional study
Record Dates: First submitted 2021-03-13; First posted 2021-03-19 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Healthy Participant
Keywords: non-carious cervical lesions; universal adhesives; smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: 47 participants having at least three non-carious cervical lesions were included in the study. Participants were divided into two groups as smokers and non-smokers. Before treatment, the dimensions and depth of the lesions were measured with periodontal probe and the sensitivity of each tooth was determined using VAS scale. All of the non-carious cervical lesions were restored with a resin composite, Essentia,GC using one of three different application modes of universal adhesive, G-Premio Bond (etch&rinse, selective-etch, self-etch). The restorations were placed by a single operator. Two calibrated examiners who were fully blind to restorative procedure evaluated the restorations in terms of retention, marginal discoloration, marginal adaptation, color match, postoperative sensitivity and secondary caries using modified USPHS criteria. The plaque and gingival index were also asessed at baseline and every 6 months of clinical service for 18 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-Premio universal adhesive used in smoker participants (Other): Participants who smoke at least 10 cigarettes per day
  Interventions: Device: G-Premio Bond in etch&rinse mode; Device: G-Premio Bond in selective-etch mode; Device: G-Premio Bond in self-etch mode
- G-Premio universal adhesive used in non-smoker participants (Other): participants who non-smoke have never smoked before
  Interventions: Device: G-Premio Bond in etch&rinse mode; Device: G-Premio Bond in selective-etch mode; Device: G-Premio Bond in self-etch mode

INTERVENTIONS:
Device: G-Premio Bond in etch&rinse mode — The phosphoric acid gel was applied to enamel and dentin washed for 5s and was dried gently with air spray. The adhesive system was applied to enamel and dentin surfaces and leave it in place for 10s.
Device: G-Premio Bond in selective-etch mode — The phosphoric acid was applied only on enamel for 10-15s then washed and was gently dried with air spray. The adhesive system was applied to enamel and dentin surfaces.
Device: G-Premio Bond in self-etch mode — The adhesive system was applied to the enamel and dentin surfaces.

SUMMARY:
The aim of the study was to evaluate the influence of smoking on the clinical performance of a universal adhesive used with different application modes in non-carious cervical lesions.

DETAILED DESCRIPTION:
Forty-seven patients (having at least three noncarious cervical lesions) were participated in this study. After allocation of patients into 2 groups according to their smoking habits (non-smokers; 24, smokers;23), lesions in each patient were restored with a resin composite, (Essentia, GC) using a universal adhesive G-Premio Bond and phosphoric acid (i-Dental) in three different application modes (etch&rinse, selective-etch or self-etch). The restorative treatments were performed by single operator. Two experienced and calibrated examiners evaluated the restorations for retention, marginal discoloration, marginal adaptation, color match, postoperative sensitivity and secondary caries at one week (baseline), at 6-, 12, and 18 months using modified USPHS criteria.While the USPHS criteria measure the clinical performance of the restorative material, it scores according to three different degrees;Alpha:The restoration is clinically perfect. Bravo:All features of the restoration are sufficient, need not be renewed. Charlie: the restoration is clinically unsuccessful, unacceptable. The gingival and plaque index were also assessed with a periodontal probe.

ELIGIBILITY:
Inclusion Criteria:

* Patients were 18 years of age or older,
* good general health,
* acceptable oral hygiene level,
* no possible health problems (such as allergies) related to resin-based restorations,
* at least three non-carious cervical lesions with at least 20 teeth in the occlusion.
* The depth of the lesions should be at least 1 mm, without carious, not previously restored, having teeth with vital, enamel and dentin tissue.
* Patients who smoke at least 10 cigarettes per day, however patients in non-smokers have never smoked before.

Exclusion Criteria:

* Participant had fewer than 20 teeth,
* having poor oral hygiene,
* uncontrolled periodontal disease,
* xerostomia,
* diagnosis of bruxism,
* pregnancy or breastfeeding possible health problems (such as allergy) related to resin-based restorations
* having severe systemic disease,
* having bleaching treatment or orthodontic treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Retention | baseline (one week)-18-month
  According to the usphs criteria, retention indicates whether a restorative material is functional in the oral environment, and is the most important criterion by which we can evaluate the success of the material.
  Alpha: Retained. Charlie: Mobile or missing; clinically unacceptable.
Marginal Discoloration | baseline (one week)-18-month
  Evaluation of color changes in restoration margins and linear staining along restoration margins. Alfa: No discoloration along the margin. Bravo: Slight and superficial staining (removable, usually localized). Charlie: Deep staining cannot be polished away.
Marginal Adaptation | baseline (one week)-18-month
  The marginal adaptation criterion evaluates the complete achievement of tooth-restoration integrity.
  Alpha: Undetectable. Bravo: Visible evidence of a crevice along the margin, dentin not exposed, clinically acceptable.
  Charlie: Explorer penetrates into crevice, dentin is exposed; clinically unacceptable.
Color match | baseline (one week)-18-month
  Evaluating whether the restoration and adjacent tooth tissue color is compatible.
  Alpha:Matches tooth. Bravo: Acceptable mismatch. Charlie:Unacceptable mismatch.
Post-op Hypersensitivity | baseline (one week)-18-month
  It is the evaluation of sensitivity after dental treatment. Alpha: Hypersensitivity absent. Charlie: Present; clinically unacceptable.
Secondary Caries | baseline (one week)-18-month
  In this criterion, the dark colored area that occurs under the tooth tissue surface and in the tooth tissue adjacent to the restoration is defined as caries.
  Alpha: Caries absent. Charlie: Present; clinically unacceptable.

SECONDARY OUTCOMES:
VAS scale | baseline (one week)-18-month
  Sensitivity to air was assessed by appling a stream of compressed air for three second 1 cm away from the tooth surface while shielding the neighboring teeth with the fingers. After this application, individuals are asked to evaluate the sensitivity of the tooth according to the Visual Analog Scale (VAS). VAS consists of a straight line 10 centimeters (cm) long. The left end of the line is 0 and it means "no pain, the right end is 10", meaning unbearable pain. With the help of this scale, the pain levels in the teeth of individuals with hypersensitivity can be determined.

OTHER OUTCOMES:
Plaque Index | baseline (one week)-18-month
  When evaluating Plaque Index scores, only the amount of plaque in the gingival area of the tooth surfaces is taken into account. Plaque amount is evaluated with periodontal probe and scored.
  Plaque Index Scores 0 When examined with a periodontal probe at the edge of the gum, no plaque accumulation is seen.
  1. When examined with a periodontal probe, it is seen that there is plaque accumulation.
  2. Visible plaque accumulation at the edge of the gum but not completely filled in the interdental area.
  3. An easily visible plaque accumulation on the gum edge and towards the coronal, completely filling the interdental zone
Gingival index | baseline (one week)-18-month
  The periodontal probe is used to evaluate whether there is inflammation, discoloration, and gingival bleeding along the gingival sulcus.
  Gingival Index Scores 0 Healthy gums.
  1. Mild inflammation: Slight discoloration and mild edema, but no bleeding on probing.
  2. Moderate inflammation: The gingiva is shiny, there is slight redness, edema and bleeding on the gum when touched with the sond.
  3. Severe inflammation: There is marked redness, edema and ulceration of the gums, the gum tends to bleed spontaneously.

CONTACTS AND LOCATIONS:
Overall Officials: A. Ruya Yazici, Principal Investigator — Study Principal Investigator
Locations (1):
- Hacettepe University Faculty of Dentistry, Ankara, Turkey (Türkiye)